CLINICAL TRIAL: NCT03780400
Title: Physical Activity Pathway for Patients With Osteoarthritis in Primary Care
Brief Title: Physical Activity Pathway for Patients With Osteoarthritis in Primary Care (OA-PCP)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Carolina, Chapel Hill (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 18-0877; 1R21AG056568 (NIH)
Record Dates: First submitted 2018-12-17; First posted 2018-12-19 (Actual); Results first posted 2020-08-25 (Actual); Last update posted 2020-08-25 (Actual); Status verified 2020-07

CONDITIONS: Osteoarthritis
Keywords: Osteoarthritis; Knee Osteoarthritis; Hip Osteoarthritis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee; Osteoarthritis, Hip

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Osteoarthritis Physical Activity Care Pathway (Experimental): 4 month physical activity (PA) counseling intervention
  Interventions: Behavioral: Osteoarthritis Physical Activity Care Pathway

INTERVENTIONS:
Behavioral: Osteoarthritis Physical Activity Care Pathway — The intervention includes brief physical activity (PA) counseling delivered via phone by a PA Counselor trained in relevant aspects of PA and motivational interviewing. During the initial call, the PA counselor will assess readiness for change in PA and will utilize appropriate PA counseling components to assess participant's PA preferences/needs, as well as referral to PA resources and goal setting. Approximately two weeks after the initial call, the PA counselor will contact participants to check in on whether they have successfully connected with PA programs or resources discussed, review progress toward PA goals and set new goals. Participants will be provided with linkage to PA programs and resources to include: self-directed, group classes/community, physical therapy and other clinical/supervised programs. Three months after the initial call, the PA counselor will call participants to assess PA and stage of change using appropriate PA counseling components and goal setting.

SUMMARY:
This is a multi-phase study that will develop and test an osteoarthritis (OA) primary care Physical activity Care Pathway (OA-PCP), a scalable intervention that includes: 1) a practical process for physical inactivity screening in primary care, 2) a brief, tailored physical activity (PA) counseling intervention via telephone, 3) connection of patients with community programs and other resources to support PA, and 4) follow-up with patients to deliver additional appropriate counseling and referrals to PA resources.

DETAILED DESCRIPTION:
This study will be a single group pilot trial of the OA-PCP. The feasibility and acceptability of the OA-PCP will be assessed among n=60 patients with hip and knee OA in two primary care clinics. All patients in the trial will participate in the OA-PCP and will complete assessments at baseline and 4-month follow-up. Feasibility metrics will include rates of recruitment, intervention engagement and retention; acceptability will be assessed from both patients and health care providers.

ELIGIBILITY:
Inclusion Criteria:

* Physician diagnosis of knee or hip OA
* Current Joint Symptoms
* Current Weekly Physical Activity <150 minutes per week.

Exclusion Criteria:

* Pain in chest when performing physical activity
* Pain in chest when not performing physical activity
* Loss of balance because of dizziness or loss of consciousness
* Recommendation from doctor to only perform physical activity under medical supervision
* No documented diagnosis of knee or hip OA
* Dementia or other memory loss condition
* Active diagnosis of psychosis
* Active Substance abuse disorder
* Total knee or hip replacement surgery, meniscus tear, ligament tear, or other significant lower extremity injury or surgery in the last 6 months
* Severe hearing or visual impairment
* Serious/terminal illness as indicated by referral to hospice or palliative care
* Unstable angina
* Hospitalization for cardiovascular event in last 6 months
* History of ventricular tachycardia
* Unstable chronic obstructive pulmonary disease (2 hospitalizations within the previous 6 months and/or on oxygen)
* Stroke with moderate to severe aphasia
* Recent history (last 6 months) of three or more falls

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 60 (Actual)
Dates: Start 2019-03-21 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kelli D Allen, PhD, Principal Investigator — UNC Chapel Hill
Locations (1):
- UNC Thurston Arthritis Research Center, Chapel Hill, North Carolina, United States

REFERENCES:
- [Derived] Beauchamp T, Arbeeva L, Cleveland RJ, Golightly YM, Hales DP, Hu DG, Allen KD. Accelerometer-Based Physical Activity Patterns and Associations With Outcomes Among Individuals With Osteoarthritis. J Clin Rheumatol. 2022 Mar 1;28(2):e415-e421. doi: 10.1097/RHU.0000000000001750. PMID 33902099
- [Derived] Allen K, Vu MB, Callahan LF, Cleveland RJ, Gilbert AL, Golightly YM, Griesemer I, Grimm K, Hales DP, Hu DG, Huffman K, Nelson AE, Pathak A, Rees J, Rethorn ZD, Wandishin AE. Osteoarthritis physical activity care pathway (OA-PCP): results of a feasibility trial. BMC Musculoskelet Disord. 2020 May 16;21(1):308. doi: 10.1186/s12891-020-03339-6. PMID 32416715

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants with symptomatic, physician diagnosed knee or hip osteoarthritis (OA) were recruited from participating primary care providers in 3 University of North Carolina clinics between March 2019 and July 2019. The first participant was enrolled on March 21, 2019 and the last participant was enrolled on July 3, 2019.
Groups:
- OA-PCP: Participants received the Osteoarthritis Physical activity Care Pathway (OA-PCP) intervention.
Period: Overall Study
Arm/Group | OA-PCP
Started | 60
Completed | 53
Not Completed | 7
Not completed — Lost to Follow-up | 5
Not completed — Withdrawal by Subject | 2

BASELINE CHARACTERISTICS:
Arm/Group | OA-PCP
Number analyzed (Participants) | 60
Age, Continuous [Mean (Standard Deviation); unit: years] | 72.4 (5.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 49
  Male | 11
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2
  Not Hispanic or Latino | 49
  Unknown or Not Reported | 9
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 1
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 15
  White | 41
  More than one race | 2
  Unknown or Not Reported | 1
Education [Count of Participants; unit: Participants] — Participants reporting at least some college.
  Participants | 48
Marital Status [Count of Participants; unit: Participants] — Participants reporting married or living with partner.
  Participants | 38
Work Status [Count of Participants; unit: Participants] — Participants reporting working full or part time.
  Participants | 17
Body Mass Index (BMI) [Mean (Standard Deviation); unit: kg/m^2] | 33.4 (7.3)
Number of Comorbid Illnesses [Mean (Standard Deviation); unit: illnesses] — Participants reported if they have or do not have these health conditions: heart disease, high blood pressure, lung disease, diabetes, ulcer/stomach diseases, kidney disease, liver disease, anemia or other blood diseases, cancer, depression, osteoarthritis/degenerative arthritis, back pain, rheumatoid arthritis or other health conditions (participant can report up to 3 other health conditions). Possible range 0 to 16.
  illnesses | 4.3 (1.7)
Years with Arthritis Symptoms [Mean (Standard Deviation); unit: years] | 11.1 (9.5)
Number of Joints with Arthritis Symptoms [Mean (Standard Deviation); unit: joints] | 7.7 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline to Month 4 for Minutes of Moderate to Vigorous Intensity PA Per Week
Description: Minutes of moderate to vigorous intensity physical activity (MVPA) per week measured via accelerometer
Time Frame: Baseline, Month 4 (Follow-up)
Population: 7 participants did not complete month 4 follow-up assessment and 11 participants had inadequate physical activity data
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | OA-PCP
Number analyzed (Participants) | 42
minutes | 0.78 [-1.6 to 3.2]
Statistical Analysis 1: Comparison: OA-PCP; Test type: Other — test for within group change from baseline to 4 month follow-up; p = 0.5145, t-test, 2 sided

2. Secondary Outcome: Change From Baseline to Month 4 for Steps Per Day
Description: Step counts were measured via an accelerometer device.
Time Frame: Baseline, Month 4 (Follow-up)
Population: 7 participants did not complete month 4 follow-up assessment and 11 participants had inadequate physical activity data
Measure: Mean (95% Confidence Interval); unit: steps
Arm/Group | OA-PCP
Number analyzed (Participants) | 42
steps | 143.7 [-174.9 to 462.2]
Statistical Analysis 1: Comparison: OA-PCP; Test type: Other — test for within group change from baseline to 4 month follow-up; p = 0.3683, t-test, 2 sided

3. Secondary Outcome: Change From Baseline to Month 4 for Minutes of Sedentary Activity
Description: Minutes of sedentary activity were measured via an accelerometer device.
Time Frame: Baseline, Month 4 (Follow-up)
Population: 7 participants did not complete month 4 follow-up assessment and 11 participants had inadequate physical activity data
Measure: Mean (95% Confidence Interval); unit: minutes
Arm/Group | OA-PCP
Number analyzed (Participants) | 42
minutes | -0.15 [-17.0 to 16.7]
Statistical Analysis 1: Comparison: OA-PCP; Test type: Other — test for within group change from baseline to 4 month follow-up; p = 0.9858, t-test, 2 sided

4. Secondary Outcome: Change From Baseline to Month 4 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Function Subscale
Description: The Western Ontario and McMasters Universities Osteoarthritis (WOMAC) function subscale includes 17 items rated on a Likert scale of 0 (no difficulty) to 4 (extreme difficulty), with ranges of 0-68 for the function subscale with higher scores indicating worse symptoms and function.
Time Frame: Baseline, Month 4 (Follow-up)
Population: 7 participants did not complete month 4 follow-up assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OA-PCP
Number analyzed (Participants) | 53
units on a scale | -6.1 [-8.7 to -3.4]
Statistical Analysis 1: Comparison: OA-PCP; Test type: Other — test for within group change from baseline to 4 month follow-up; p < 0.0001, t-test, 2 sided

5. Secondary Outcome: Change From Baseline to Month 4 in Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Pain Subscale
Description: The Western Ontario and McMasters Universities Osteoarthritis (WOMAC) Pain Subscale is a measure of lower extremity pain. It includes 5 items rated on a Likert scale of 0 (no pain) to 4 (extreme pain), with a total range of 0-20 with higher scores indicating worse symptoms and function.
Time Frame: Baseline, Month 4 (Follow-up)
Population: 7 participants did not complete month 4 follow-up assessment
Measure: Mean (95% Confidence Interval); unit: units on a scale
Arm/Group | OA-PCP
Number analyzed (Participants) | 53
units on a scale | -1.9 [-2.7 to -1.0]
Statistical Analysis 1: Comparison: OA-PCP; Test type: Other — test for within group change from baseline to 4 month follow-up; p < 0.0001, t-test, 2 sided

ADVERSE EVENTS:
Time Frame: Data was collected starting at baseline to 4 months, ending at participants' final follow up time point.
Arm/Group | OA-PCP
All-Cause Mortality (participants affected / at risk) | 0/60
Serious Adverse Events (participants affected / at risk) | 0/60
Other Adverse Events (participants affected / at risk) | 0/60

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-07-01): https://cdn.clinicaltrials.gov/large-docs/00/NCT03780400/Prot_SAP_000.pdf